CLINICAL TRIAL: NCT02323321
Title: International Trial to Evaluate the Safety and Effectiveness of The Portable Organ Care System (OCS™) Heart For Preserving and Assessing Expanded Criteria Donor Hearts for Transplantation (EXPAND Heart Trial)
Brief Title: International EXPAND Heart Pivotal Trial
Acronym: EXPANDHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-CAR-012014
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2019-08

CONDITIONS: Heart Transplant
Keywords: heart transplant; heart preservation; beating heart transplant
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCS Preservation (Experimental): OCS Preservation and Assessment
  Interventions: Device: Preservation of Hearts for Transplantation

INTERVENTIONS:
Device: Preservation of Hearts for Transplantation — Preserving and Assessing Expanded Criteria Donor Hearts for Transplantation

SUMMARY:
To evaluate the effectiveness of the OCS™ Heart to recruit, preserve and assess donor hearts that may not meet current standard donor heart acceptance criteria (as identified above) for transplantation to potentially improve donor heart utilization for transplantation

ELIGIBILITY:
Inclusion Criteria:

* Registered male or female primary Heart transplant candidate
* Age ≥18 years old

Exclusion Criteria:

* Prior solid organ or bone marrow transplant
* Chronic use of hemodialysis or diagnosis of chronic renal insufficiency
* Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2019-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCS Preservation
Started | 75
Completed (Completed one-year follow-up) | 62
Not Completed | 13
Not completed — Re-Transplant | 1
Not completed — Death | 12

BASELINE CHARACTERISTICS:
Groups:
- OCS Preservation: OCS Heart System: The OCS Heart System preserves the heart in a near-physiological, beating state by perfusing the heart with a warmed, donor-blood based perfusate that is supplemented with nutrients and oxygen in a controlled and protected environment
Arm/Group | OCS Preservation
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.46 (12.556)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 58
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival at Day-30 Post Transplant and Absence of Severe Primary Heart Graft Dysfunction in the First 24 Hours Post-transplantation
Description: A composite endpoint of patient survival at Day-30 post-transplant and absence of severe heart primary graft dysfunction (PGD) (left or right ventricle)) in the first 24 hours post-transplantation.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Preservation
Number analyzed (Participants) | 75
Participants | 66
Statistical Analysis 1: Comparison: OCS Preservation; Test type: Other — The primary hypothesis for this study is that the true (success) proportion of transplanted patients meeting the primary effectiveness endpoint, patient survival at day 30 post-transplantation and absence of severe PGD (left or right ventricle) in the first 24 hours post-transplantation, is greater than the Performance Goal value of 0.65; p < 0.0001, one-sided exact binomial test; Proportion = 88.0, 95% CI 2-sided [78.4 to 94.4]

ADVERSE EVENTS:
Time Frame: Per the protocol, all SAEs and heart graft related SAEs will be collected for the first 30 days post-transplant. All-Cause Mortality was assessed for 12 months post-transplant as reported.
Description: Per the protocol, only serious adverse events (SAEs) and Heart Graft-Related SAE's (HGRSAEs) will be captured in this study.
  Not Serious AEs were not collected, and therefore not reported.
Arm/Group | OCS Preservation
All-Cause Mortality (participants affected / at risk) | 12/75
Serious Adverse Events (participants affected / at risk) | 56/75
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Preservation (N=75)
Arrhythmia (Cardiac disorders) | 4 (4)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Cor pulmonale (Cardiac disorders) | 2 (2)
Electromechanical dissociation (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 5 (5)
Left ventricular failure (Cardiac disorders) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 5 (5)
Right ventricular dysfunction (Cardiac disorders) | 4 (4)
Right ventricular failure (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Heart transplant rejection (Immune system disorders) | 12 (12)
Clostridial infection (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 3 (3)
Heart injury (Injury, poisoning and procedural complications) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Rectal laceration postoperative (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 10 (10)
Renal impairment (Renal and urinary disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Haemorrhage (Vascular disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02323321/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02323321/SAP_001.pdf